CLINICAL TRIAL: NCT05303389
Title: Posterior Plating Versus Anterior to Posterior Screws in Fixation of Posterior Column in Pilon Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M D 193 / 2020
Record Dates: First submitted 2022-03-10; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Tibial Fractures
MeSH Terms: conditions — Tibial Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Posterior plating group (Experimental): Fix the posterior fragment using a buttress plate through a posterolateral approach by an interval between flexor hallucis longus and peroneii.
  Interventions: Procedure: Fixation of 2,3 or 4 column pilon fracture of the tibia
- Anterior to posterior group (Active Comparator): Fix the posterior fragment using anterior to posterior 4.0 mm cannulated screws under xray guidance.
  Interventions: Procedure: Fixation of 2,3 or 4 column pilon fracture of the tibia

INTERVENTIONS:
Procedure: Fixation of 2,3 or 4 column pilon fracture of the tibia — anterior to posterior screws in classic arm and posterolateral approach in new arm group

SUMMARY:
Management of comminuted distal tibia fracture (pilon fracture) is still a challenging field. It is recently done guided by the new four column theory of distal tibia. Several approaches were advocated to address and fix each column. Fixation of posterior column is still a wide debate among orthopedic surgeons. This study is conducted to compare outcomes between two modalities for the management of posterior column fracture in pilon fractures.

DETAILED DESCRIPTION:
The aim of this work is to assess and compare results of anterior to posterior screws versus posterior buttress plate in management of posterior column fracture in pilon fracture as regards functional, radiological outcomes and possible complications.

Optimal treatment of comminuted pilon fractures requires precise anatomical reduction. Several methods have been advocated to manage complex pilon fractures, but an optimal fixation technique remains controversial. On the basis of the anatomical characteristics of the ankle joint a four-column classification to guide the treatment of comminuted pilon fractures was proposed. The four-column classification can be summarized as follows: lateral column( the distal fibula), posterior column( the posterior part of the intermalleolus line with the distal tibial shaft), anterior column (the anterior part of the intermalleolus line with the distal tibial shaft) and medial column(the medial one-third of the tibial plafond with the distal tibial shaft).

A posterolateral incision is typically used to reduce and fix the posterior malleolar fragment to the tibial metaphysis which can be also done through the anterior incision using anterior to posterior screws.

ELIGIBILITY:
Inclusion Criteria:

* Two, Three and four column pilon fracture

Exclusion Criteria:

* Pathological fractures.
* Pediatric age group with open physis.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
The American Orthopaedic Foot and Ankle Society (AOFAS) scoring system | up to one year
  A system measuring function, alignment and pain in the operated ankle. The score maximum is 100 points, where a higher score indicates better recovery .

CONTACTS AND LOCATIONS:
Overall Officials: Tamer Fayyad, MD, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baraka MM, Fayyad TA, Thakeb MF, Lamei MA, Al Kersh MA. Posterior Plating Versus Anterior to Posterior Screws in Fixation of Posterior Column in Pilon Fractures. J Orthop Trauma. 2025 Jun 1;39(6):288-295. doi: 10.1097/BOT.0000000000002966. PMID 39976678